CLINICAL TRIAL: NCT06954987
Title: A Two Cohort, Randomized, Double-Blind, Placebo-Controlled, Phase II Multi-Center Signal-Finding Study of Venetoclax Combined With Reduced-Intensity Conditioning Followed by Allogeneic Hematopoietic Cell Transplantation Then Venetoclax Maintenance in Adult Patients With Acute Myeloid Leukemia in First Complete Remission: A MyeloMATCH Sub-Study
Brief Title: Venetoclax or Placebo in Combination With Reduced-Intensity Conditioning Hematopoietic Cell (Bone Marrow/Blood Stem Cell) Transplant and as Maintenance Therapy After Transplant in Patients With Acute Myeloid Leukemia (A MyeloMATCH Treatment Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2025-03015; NCI-2025-03015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM3TCT-A03 (Other: Alliance for Clinical Trials in Oncology); MM3TCT-A03 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2025-05-01; First posted 2025-05-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Busulfan; X-Rays; fludarabine; Melphalan; Magnetic Resonance Spectroscopy; Whole-Body Irradiation; venetoclax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, double-blind trial. Sites will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Conditioning 1A (matched donors with venetoclax) (Experimental): Patients receive venetoclax PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Busulfan; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Venetoclax
- Conditioning 1B (matched donor with placebo) (Placebo Comparator): Patients receive placebo PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Busulfan; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Placebo Administration; Procedure: Positron Emission Tomography
- Conditioning 2A (haplo/mismatched donor with venetoclax) (Experimental): Patients receive venetoclax PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Radiation: Total-Body Irradiation; Drug: Venetoclax
- Conditioning 2B (haplo/mismatched unrelated and placebo) (Placebo Comparator): Patients receive placebo PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Placebo Administration; Procedure: Positron Emission Tomography; Radiation: Total-Body Irradiation
- Maintenance I (venetoclax) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Drug: Venetoclax
- Maintenance II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Placebo Administration; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Given IV
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Procedure: Biospecimen Collection — Undergo blood, urine and buccal swab collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo)
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 1B (matched donor with placebo); Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Drug: Placebo Administration — Given PO
  Arms: Conditioning 1B (matched donor with placebo); Conditioning 2B (haplo/mismatched unrelated and placebo); Maintenance II (placebo)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Total-Body Irradiation — Undergo total body irradiation
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
  Arms: Conditioning 2A (haplo/mismatched donor with venetoclax); Conditioning 2B (haplo/mismatched unrelated and placebo)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Conditioning 1A (matched donors with venetoclax); Conditioning 2A (haplo/mismatched donor with venetoclax); Maintenance I (venetoclax)

SUMMARY:
This phase II MyeloMATCH treatment trial compares the effect of adding venetoclax or placebo to reduced intensity conditioning chemotherapy with fludarabine and busulfan or melphalan, with or without total body irradiation, followed by hematopoietic stem cell transplant and either venetoclax or placebo maintenance therapy after transplant, for the treatment of patients with acute myeloid leukemia (AML). Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving chemotherapy and total body irradiation before a donor stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells. Adding venetoclax to conditioning therapy before, and giving it as maintenance therapy after, a hematopoietic stem cell transplant may be a more effective treatment option than the usual approach in patients with AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if venetoclax combined with reduced-intensity conditioned allogeneic hematopoietic cell transplantation improves 100-day event-free survival relative to placebo in adults with AML in first complete remission (complete remission [CR] or complete remission with incomplete hematologic recovery [CRi]).

SECONDARY OBJECTIVES:

I. To determine the post-transplant 30-day and 12-month event-free survival (EFS) rates in venetoclax and placebo arms.

II. To determine the post-transplant 12-month EFS in patients with minimal/measurable residual disease (MRD)-positive status first complete remission at transplant in venetoclax and placebo arms.

III. To determine the post-transplant 100-day and 12-month overall survival (OS) rate in venetoclax and placebo arms.

IV. To determine the post-transplant 100-day and 12-month cumulative incidence rates (CIR) of morphologic relapse in venetoclax and placebo arms.

V. To determine the post-transplant 100-day and 12-month non-relapse mortality (NRM) rates in venetoclax and placebo arms.

VI. To determine the post-transplant 12-month relapse-free survival rate (RFS), OS, cumulative incidence of relapse (CIR), and cumulative incidence of NRM from start of maintenance in venetoclax and placebo arms.

VII. To determine the post-transplant 100-day and 12-month cumulative incidence of grade 2-4 acute graft versus host disease (GVHD) and 12-month cumulative incidence of chronic GVHD.

VIII. To determine neutrophil engraftment at day 30 and platelet engraftment at days 30 and 60 post-transplant.

IX. To determine the incidence of primary and secondary graft failure within 12 months of hematopoietic stem cell transplant (HCT).

X. To assess toxicity and tolerability of the combination of reduced intensity conditioned allogeneic hematopoietic cell transplantation and venetoclax.

EXPLORATORY OBJECTIVES:

I. To determine the post-transplant 30-day MRD clearance rates in venetoclax and placebo arms.

II. To assess patterns of immune reconstitution per standard of care (SOC) site testing for venetoclax and placebo arms.

III. To assess patterns of marrow and peripheral blood chimerism per SOC site testing for venetoclax and placebo arms.

IV. To assess graft-versus-host relapse-free survival for venetoclax and placebo arms.

V. To assess clinical flow and genetic MRD concordance rate (using Myelomatch available MRD tools) and to associate MRD negativity with clinical outcomes for venetoclax and placebo arms.

VI. Compare rate of cytokine release syndrome after hematopoietic cell infusion. (Cohort 2 only)

OUTLINE: Patients with matched donors are randomized to conditioning 1A or 1B. Patients with haploidentical or mismatched unrelated donors are randomized to conditioning 2A or 2B.

CONDITIONING 1A: Patients receive venetoclax orally (PO) once daily (QD) on days -10 to -2, fludarabine intravenously (IV) on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or twice daily (BID) on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 1B: Patients receive placebo PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 2A: Patients receive venetoclax PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 2B: Patients receive placebo PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: All patients without evidence of relapse at day +100 are re-randomized to maintenance I or II.

MAINTENANCE I: Patients receive venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE II: Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity.

Patients undergo chest x-ray, echocardiography or multigated acquisition scan (MUGA) during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo positron emission tomography (PET) scan and/or computed tomography (CT) scan throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3 months for up to 1 year and then every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be registered to the Master Screening and Reassessment Protocol (MSRP) and assigned to this protocol by the MATCHBox Treatment Verification Team
* STEP 1: History of acute myeloid leukemia (AML) by World Health Organization (WHO) criteria in first complete remission with morphologic complete remission (CR) or CR with incomplete hematologic recovery (CRi) defined as less than 5% bone marrow blasts by morphology with no circulating leukemic myeloblasts and no known extramedullary disease
* STEP 1: MRD status by MDNet must have been performed
* STEP 1 COHORT 1: Human leukocyte antigen (HLA)-matched donor defined as one of the following:

  * Sibling donor must be a 6/6 match at HLA-A and -B (intermediate or higher resolution) and -DRB1 (at high resolution using deoxyribonucleic acid [DNA]-based typing)
  * Related donor other than sibling must be an 8/8 match for HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing
  * Unrelated donor must be an 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing
  * Age 40-75 years
* STEP 1 COHORT 1: Not recommended for a myeloablative regimen by treating investigator
* STEP 1 COHORT 2: Haploidentical or HLA-mismatched unrelated donor defined as one of the following:

  * Haploidentical donors: Related donor must be a haploidentical 3/6, 4/6, or 5/6 match at HLA-A and -B (intermediate or higher resolution) and -DRB1 (at high resolution using DNA-based typing)
  * HLA-mismatched unrelated donors: Unrelated donor must be a 6/8 or 7/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing, ideally age < 35
  * Age 18-75 years
* STEP 1 COHORT 2: Not recommended for a myeloablative regimen by treating investigator
* STEP 1: Prior venetoclax therapy is allowed unless there is evidence of progression or no response (failure to achieve remission) to venetoclax-based regimen < 2 months prior to registration
* STEP 1: No prior allogeneic or autologous hematopoietic cell transplantation
* STEP 1: Anti-leukemic therapy must be completed more than 14 days prior to registration with the exception of venetoclax
* STEP 1: Karnofsky performance status ≥ 60
* STEP 1: Total bilirubin < 2 x upper limit of normal (ULN)
* STEP 1: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 3 x upper limit of normal (ULN)
* STEP 1: Alkaline phosphatase ≤ 2.5 x upper limit of normal (ULN)
* STEP 1: Pulmonary function diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) ≥ 40% and forced expiratory volume (FEV1) ≥ 50%
* STEP 1: Calculated (Calc.) creatinine clearance ≥ 40 mL/min/based on the Cockcroft-Gault formula
* STEP 1: Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done ≤ 7 days prior to registration is required
* STEP 1: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* STEP 1: Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* STEP 1: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* STEP 1: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* STEP 1: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. To be eligible for this trial, patients should have ejection fraction ≥ 40% and NYHA functional status class II or better
* STEP 1: No history of liver cirrhosis
* STEP 1: No history of sinusoidal occlusion syndrome of the liver
* STEP 1: No known intolerance or allergy to any protocol-defined agents
* STEP 1: No known medical condition causing an inability to swallow oral formulations of agents
* STEP 2: Patient has completed the conditioning and transplantation regimens
* STEP 2: Patient has no evidence of AML morphologic relapse
* STEP 2: Patient does not have flow measurable/minimal residual disease by myeloMATCH central labs (MDNet) testing defined as ≥ 0.1% on day 100+ (between day 80+ and 110+) marrow
* STEP 2: Absolute neutrophil count > 1,000/mcL (confirmed by a lab draw performed on two separate occasions [> 2 days apart])
* STEP 2: Platelet count > 50,000/mcL
* STEP 2: AST (SGOT)/ALT (SGPT) < 3 x upper limit of normal (ULN)
* STEP 2: Total bilirubin < 2 mg/dL x upper limit of normal (ULN)
* STEP 2: Calc. creatinine clearance ≥ 40 mL/min/based on the Cockcroft-Gault formula
* STEP 2: Patient does not have active/current grade 3-4 acute GVHD
* STEP 2: Patient does not have evidence of grade 3 or higher sinusoidal occlusion syndrome/veno-occlusive disease of the liver as defined by European Society for Blood and Marrow Transplantation (EBMT) criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2026-03-18 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | From randomization to minimal residual disease (MRD) persistence, MRD relapse, morphologic relapse, or death from any cause, assessed up to day +100
  MRD positivity is defined as >= 0.1% leukemic blasts by MyeloMatch flow cytometry. Day 100 is defined as 100 days (day +100 +/- 10 days) after hematopoietic cell infusion (day 0). The day 100 EFS rates will be compared between venetoclax versus placebo arms using a using a two-sided log-rank test.

SECONDARY OUTCOMES:
MRD conversion rate | At day +30
  Corresponding 95% binomial confidence intervals will be estimated at 30 days. Proportions will be compared using Fisher's test or Chi-square test. The analysis will be done within each cohort.
EFS | From the time of randomization to relapse or death, assessed at 12 months
  Kaplan-Meier estimates and their corresponding 95% binomial confidence intervals will be estimated at 12 months. The analysis will be done within each cohort.
Overall survival | From randomization to death from any cause, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method for each treatment.
Relapse free survival | From randomization or re-randomization to morphologic relapse or death from any cause, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method for each treatment.
Non relapse mortality | From randomization to death from any cause other than morphologic relapse, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method for each treatment.
Cumulative incidence of morphologic relapse | From the date of achievement of a remission until the date morphologic relapse, assessed up to 10 years
Incidence of acute graft versus host disease (GVHD) | From date of randomization until date of death with acute GVHD
  Gray's test was used to assess the difference between venetoclax and placebo arms.
Incidence of chronic GVHD | From date of randomization until date of death with chronic GVHD
  Gray's test was used to assess the difference between venetoclax and placebo arms.
Time of neutrophil engraftment | Up to 10 years
  Defined as the first of three successive days with absolute neutrophil count ≥ 0.5 × 10^9/L after post-transplantation nadir.
Time of platelet engraftment | Up to 10 years
  Defined as the first of seven consecutive days with platelet count 20 × 10^9/L or higher, in the absence of platelet transfusion for preceding seven days.
Incidence of adverse events | Up to 10 years
  Frequency and severity of adverse events and tolerability for each treatment strategy group will be summarized using descriptive statistics. As per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, the term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. Will also assess tolerability through assessing the number of patients who require dose modifications and/or dose delays, and the proportion of patients who go off treatment due to adverse events. Further, toxicity and tolerability measures will be assessed by treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Wieduwilt, Principal Investigator — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm